CLINICAL TRIAL: NCT01035190
Title: Efficacy and Safety of Inhaled Budesonide in Very Preterm Infants at Risk for Bronchopulmonary Dysplasia
Acronym: NEuroSIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Children's Hospital Tuebingen (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Dirk Bassler, Msc, Prof.Dr. med., University Children's Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GAH-F5_2009-223060
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Preterm Infants; Inhaled Corticosteroids; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- inhaled Budesonide (Experimental)
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Inhalation, 200 µg/puff
  Other Names: Budiair

SUMMARY:
HYPOTHESIS:

Early prophylactic inhalation of Budesonide reduces the absolute risk of developing bronchopulmonary dysplasia (BPD) or death in preterm infants born <28 weeks gestational age (GA) by 10%.

PRIMARY OBJECTIVE:

To determine whether inhalation of Budesonide within 12 hours of life improves survival without BPD at 36 weeks GA in infants born between 23 and 27 weeks GA.

SECONDARY OBJECTIVES:

To determine whether prophylactic inhalation of Budesonide affects neurodevelopment at a corrected age of 18-22 months in preterm infants; to determine whether inhalation of corticosteroids is associated with adverse treatment effects, alters mortality at 36 weeks GA, BPD incidence at 36 weeks GA, and the duration of positive pressure respiratory support or supplemental oxygen.

RATIONALE:

Pre- and postnatal exposure of the developing lung to inflammation is central to the development of BPD and the pulmonary inflammatory response in preterms at risk of developing BPD is established very early in life. Corticosteroids have antiinflammatory properties and early inhalation of corticosteroids may allow for beneficial local effects on the pulmonary system prior to the development of a full inflammatory response with a lower risk of undesirable systemic side effects.

STUDY DESIGN:

Randomised placebo-controlled, multi-centre clinical trial.

RESEARCH PLAN:

Within 2 years 850 infants of 23-27 weeks GA will be randomised during the first 12 hours of life to Budesonide or placebo to prevent BPD. Study drugs will be administered via Aerochamber and continued until infants are either off supplementary oxygen and positive pressure support or have reached a GA of 32 0/7 weeks regardless of ventilatory status. The primary outcome of survival without BPD will be determined at 36 weeks GA and BPD will be defined according to the physiological definition. Study patients will be followed and neurodevelopmental outcomes will be assessed at a corrected age of 18-22 months.

CLINICAL SIGNIFICANCE:

BPD not only contributes to the mortality of preterm infants but is also associated with impaired neurosensory development in Extremely Low Birth Weight (ELBW) survivors, frequent readmission to hospital in the first 2 years of life, as well as with an increased risk of asthma, lung function abnormalities and persistent respiratory symptoms in adolescence and young adulthood. Systemic corticosteroids are effective in preventing BPD, but their use is practically prohibited given their adverse effects on neurodevelopment. Early inhalation of corticosteroids has been shown to be associated with secondary pulmonary benefits, but its effect on survival without BPD and on neurodevelopment remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* a gestational age of 23 0/7-27 6/7 weeks,
* a postnatal age < 12 hours
* the necessity for any form of positive pressure support (mechanical or nasal ventilation or CPAP

Exclusion Criteria:

* involve a clinical decision not to administer therapies (infant not considered viable)
* dysmorphic features or congenital malformations that adversely affect life expectancy or neurodevelopment and known or suspected congenital heart disease

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 863 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Survival without BPD at 36 weeks GA | 36 weeks GA

SECONDARY OUTCOMES:
Neurodevelopment at a corrected age of 18 - 22 months. | 18 - 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Dirk Bassler, MSc, Principal Investigator — University Children's Hospital Tuebingen / University Hospital Zurich, Department of Neonatology; Prof. Dr. med. Christian F Poets, Principal Investigator — Children's Hospital, Tuebingen
Locations (40):
- Belgium (4):
  - AZ Sint-Jan Brugge Oostende AV, Department of Neontalogy, Bruges
  - CHU St-Pierre, UMC St-Pieter, Brussels
  - HUDERF, Department of Neonatology, Brussels
  - CHU Tivoli, Department of Neonatology, La Louvière
- Czechia (6):
  - University Hospital Brno, Department of Neonatology, Brno
  - University Hospital Ostrava, Department of Neonatology, Ostrava
  - University Hospital Plzen, Department of Neonatology, Pilsen
  - Charles University, General Faculty Hospital and 1st Faculty of Medicine, Department of Obstetrics and Gynecology, Prague
  - University Hospital Motol Prague 5, Department of Neonatology, Prague
  - University Hospital of Tomas Bati, Department of Neonatology, Zlín
- Finland (5):
  - Helsinki University Central Hospital,Hospital for Children and Adolescents, NICU, Helsinki
  - University Hospital Kuopio, NICU, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospita, NICU, Tampere
  - Tartu University Children's Clinic, Paediatric Intensive Care Unit, Tartu
- France (3):
  - CHU de LilleHôpital Jeanne de Flandres, Pôle de Médecine néonataleUnité de Réanimation néonatale, Lille
  - Hospital Cochin Saint-Vincent de Paul, Dept. of Neonatology, Paris
  - Hôpital Clocheville, Service de RéanimationNéonatale, Tours
- Germany (11):
  - University Children's Hospital Aachen, Dept. of Neonatology, Aachen
  - University Children's Hospital Carl Gustav Carus Dresden, Dept. of Neonatology, Dresden
  - University Children's Hospital Erlangen, Dept. of Neonatology, Erlangen
  - University Children's Hospital Essen, Dept. of Pediatrics, Essen
  - Georg-August University Hospital Goettingen, Dept. of Pediatrics, Göttingen
  - University Hospital Hamburg-Eppendorf, Dept. of Neonatology, Hamburg
  - Children's Hospital Hannover auf der Bult, Dept. of Neonatology, Hanover
  - University Hospital Hannover, Dept. of Neonatology, Hanover
  - University Children's Hospital Heidelberg, Dept. of Neonatology, Heidelberg
  - Hospital Nuernberg Sued, Dept. of Neonatology, Nuremberg
  - University Children´s Hospital Tuebingen, Dept. of Neonatology, Tübingen
- Israel (5):
  - Ben-Gurion University of NegevSoroka Medical Center, Neonatal Department, Beersheba
  - Bnai Zion Medical Center Haifa, Department of Neonatology, Haifa
  - Hadassah Medical Center, Department of Neonatology, Jerusalem
  - Meir Medical Center, Premature Baby Unit, Kfar Saba
  - Kaplan Medical Center Rehovot, Dept. of Neonatology, Rehovot
- Italy (5):
  - Ospedale Salesi, SOD Neonatologia, Ancona
  - ASO S. Croce e Carie, Terapia Intensiva Neonatale-Neonatologia, Cuneo
  - Azienda Ospedaliera di Padova, Dipartimento di Pediatria Salus Pueri, Padua
  - Azienda Ospedaliera Universitaria Pisana, U.O. Neonatologia, Pisa
  - Ospedale Sant'Anna, Terapia Intensiva Neonatale Clinica -3°piano, Torino
- Erasmus MC - Sophia, Department of Neonatology, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bassler D, Halliday HL, Plavka R, Hallman M, Shinwell ES, Jarreau PH, Carnielli V, van den Anker J, Schwab M, Poets CF. The Neonatal European Study of Inhaled Steroids (NEUROSIS): an eu-funded international randomised controlled trial in preterm infants. Neonatology. 2010;97(1):52-5. doi: 10.1159/000227294. Epub 2009 Jul 7. No abstract available. PMID 19590247
- [Derived] Ciora OA, Seegmuller T, Fischer JS, Wirth T, Hafner F, Stoecklein S, Flemmer AW, Forster K, Kindt A, Bassler D, Poets CF, Ahmidi N, Hilgendorff A. Delineating morbidity patterns in preterm infants at near-term age using a data-driven approach. BMC Pediatr. 2024 Apr 11;24(1):249. doi: 10.1186/s12887-024-04702-5. PMID 38605404
- [Derived] Bassler D, Shinwell ES, Hallman M, Jarreau PH, Plavka R, Carnielli V, Meisner C, Engel C, Koch A, Kreutzer K, van den Anker JN, Schwab M, Halliday HL, Poets CF; Neonatal European Study of Inhaled Steroids Trial Group. Long-Term Effects of Inhaled Budesonide for Bronchopulmonary Dysplasia. N Engl J Med. 2018 Jan 11;378(2):148-157. doi: 10.1056/NEJMoa1708831. PMID 29320647
- [Derived] Bassler D, Plavka R, Shinwell ES, Hallman M, Jarreau PH, Carnielli V, Van den Anker JN, Meisner C, Engel C, Schwab M, Halliday HL, Poets CF; NEUROSIS Trial Group. Early Inhaled Budesonide for the Prevention of Bronchopulmonary Dysplasia. N Engl J Med. 2015 Oct 15;373(16):1497-506. doi: 10.1056/NEJMoa1501917. PMID 26465983